CLINICAL TRIAL: NCT02036060
Title: Abiraterone Acetate Maintenance in Combination With Docetaxel After Disease Progression to Abiraterone Acetate in Metastatic Castration Resistant Prostate Cancer. Randomized Phase II Study.
Brief Title: Abiraterone Acetate in Combination With Docetaxel After Disease Progression to Abiraterone Acetate in Metastatic Castration Resistant Prostate Cancer.
Acronym: ABIDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Janssen, LP (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABIDO-SOGUG; 2013-003811-23 (EudraCT Number)
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic prostate cancer; Abiraterone acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; abiraterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): docetaxel 75 mg/m2 + prednisone 10 mg/d + abiraterone 1000 mg/d
  Interventions: Drug: docetaxel 75 mg/m2 + prednisone 10 mg/d + abiraterone 1000 mg/d
- Arm B (Active Comparator): docetaxel 75 mg/m2 + prednisone 10 mg/d
  Interventions: Drug: docetaxel 75 mg/m2 + prednisone 10 mg/d

INTERVENTIONS:
Drug: docetaxel 75 mg/m2 + prednisone 10 mg/d + abiraterone 1000 mg/d — Docetaxel 75 mg/m2 + prednisone 10 mg/d + abiraterone 1000 mg/d in 21 day cycles.
  Other Names: Arm A
  Arms: Arm A
Drug: docetaxel 75 mg/m2 + prednisone 10 mg/d — Docetaxel 75 mg/m2 plus prednisone 10 mg/d in 21 day cycles.
  Other Names: Arm B
  Arms: Arm B

SUMMARY:
Prostate cancer is the most frequently diagnosed non-skin cancer, and the second leading cause of men cancer death in the United States. Hormonal therapy remains a first-line treatment for metastatic prostate cancer. Initial responses to hormonal therapy with chemical or surgical castration are quite favorable, however, most patients will progress to a castration-resistant phase of the disease. Docetaxel is the primary chemotherapeutic option for patients with mCRPC.

Abiraterone is a novel, selective, irreversible, and potent inhibitor of 17-[alpha]-hydroxylase/17,20-lyase (CYP17) enzymatic activity that has recently been demonstrated to further reduce testosterone levels in the blood to undetectable range (< 1 ng/dL) and is suggested to reduce de novo intratumor androgen synthesis. Abiraterone demonstrated activity in castration resistant prostate cancer patients previously treated with docetaxel chemotherapy. Recently, results of a phase III trial comparing abiraterone plus prednisone vs placebo plus prednisone in asymptomatic and without visceral metastasis, castration-resistant metastatic prostate cancer patients, demonstrated a better radiological progression free survival for abiraterone treated patients and a trend towards a better survival was clear for abiraterone treated patients.

No clinical evidence exists about efficacy of chemotherapy and antiandrogen therapy combination. All trials have been performed in patients in which LHRH agonist treatment was continued although there is not clear evidence about efficacy of hormonal treatment. Some retrospective studies suggest that androgen deprivation treatment should be maintained in chemotherapy treated patients. Abiraterone has been proved to suppress androgen levels to negative values, and to add efficacy to castration hormonal therapy. Combination of abiraterone with docetaxel chemotherapy seems promising adding efficacy to only docetaxel chemotherapy. A randomized phase II study comparing docetaxel + prednisone + abiraterone to docetaxel + prednisone in mCRPC in patients treated previously with abiraterone, seems promising to explore addition of efficacy to taxotere after abiraterone hormonal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Male aged 18 years and above
* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Metastatic disease documented by positive bone scan or metastatic lesions other than liver or visceral metastasis on CT, MRI.
* Prostate cancer progression to previous castration treatment documented by PSA according to PCWG2 or radiographic progression according to modified RECIST criteria or bone scan progression
* Asymptomatic or mildly symptomatic from prostate cancer
* Surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 2.0 nM).
* Previous anti-androgen therapy and progression after withdrawal.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Hemoglobin >= 10.0 g/dL independent of transfusion
* Platelet count >= 100,000/µL
* Serum albumin >= 3.5 g/dL
* Serum creatinine < 1.5 x ULN or a calculated creatinine clearance >= 60 mL/min
* Serum potassium >= 3.5 mmol/L
* Liver function: a. Serum bilirubin < 1.5 x ULN (except for patients with documented Gilbert's disease) b. AST or ALT < 2.5 x ULN
* Life expectancy of at least 6 months
* Patients who have partners of childbearing potential must be willing to use a method of birth control

Exclusion Criteria:

* Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
* Any chronic medical condition requiring a higher dose of corticosteroid than 10mg prednisone/prednisolone daily.
* Pathological finding consistent with small cell carcinoma of the prostate
* Liver or visceral organ metastasis
* Known brain metastasis
* Use of opiate analgesics for cancer-related pain, including codeine and dextropropoxyphene, currently or anytime within 4 weeks of Cycle 1 Day 1
* Prior cytotoxic chemotherapy or biologic therapy for the treatment of CRPC
* Radiation therapy for treatment of the primary tumor within 6 weeks of Cycle 1, Day
* Radiation or radionuclide therapy for treatment of metastatic CRPC
* Previously treated with ketoconazole for prostate cancer for greater than 7 days
* Prior systemic treatment with an azole drug (e.g. fluconazole, itraconazole) within 4 weeks of Cycle 1, Day 1
* Prior flutamide (Eulexin) treatment within 4 weeks of Cycle 1, Day 1
* Bicalutamide (Casodex), nilutamide (Nilandron) within 6 weeks of Cycle 1 Day 1
* Uncontrolled hypertension (systolic BP >= 160 mmHg or diastolic BP >= 95 mmHg).
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease
* Atrial Fibrillation, or other cardiac arrhythmia requiring therapy
* Other malignancy, except non-melanoma skin cancer, with a >= 30% probability of recurrence within 24 months
* Administration of an investigational therapeutic within 30 days of Cycle 1, Day 1
* Any condition which, in the opinion of the investigator, would preclude participation in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-02-07 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
1 year radiologic progression free survival | 1 year
  Time from randomization to radiologic disease progression

SECONDARY OUTCOMES:
Overall survival | Up to 3 years
  Time from randomization to death
Radiologic progression free survival | Up to 1 year
  Time from randomization to radiologic progression free survival
PSA progression free survival | Up to 3 weeks
  Time from randomization to PSA progression
PSA response rate | Up to 3 weeks
  50% & 90% PSA reduction from randomisation
Objective response rate | Up to 12 weeks
  Response according RECIST criteria
Quality of life rate | Up to 12 weeks
  Quality of life according to FACT-P questionaire
Time to skeletal-related event | Up to 12 weeks
  Time from randomization to skeletal-related events
Time to opiate use for cancer pain | Up to 3 weeks
  Time from randomization to opiate use for cancer pain
Time to pain progression | Up to 3 weeks
  Time from randomization to pain progression defined as an increase in median BPI score ≥ 30% from baseline
Safety profile | Up to 3 weeks
  Related adverse events per patient

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Climent, MD, Study Chair — Fundación Instituto Valenciano de Oncología; José A Arranz, MD, Principal Investigator — HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑÓN, Servicio de Oncología Médica; Daniel E Castellano, MD, Principal Investigator — HOSPITAL UNIVERSITARIO 12 DE OCTUBRE,Servicio de Oncología Médica; Begoña Mellado, MD, Principal Investigator — HOSPITAL CLINIC I PROVINCIAL DE BARCELONA, Servicio de Oncología Médica; Albert Font, MD, Principal Investigator — HOSPITAL UNIVERSITARI GERMANS TRIAS I PUJOL, Servicio de Oncología Médica; Alfredo Sánchez, MD, Principal Investigator — CONSORCIO HOSPITALARIO PROVINCIAL DE CASTELLÓN, Servicio de Oncología Médica; Emilio Esteban, MD, Principal Investigator — HOSPITAL UNIVERSITARIO CENTRAL DE ASTURIAS, Servicio de Oncología Médica; María I Sáez, MD, Principal Investigator — HOSPITAL VIRGEN DE LA VICTORIA, Servicio de Oncología Médica; Carmen Santander, MD, Principal Investigator — HOSPITAL UNIVERSITARIO MIGUEL SERVET, Servicio de Oncología Médica; Pablo Maroto, MD, Principal Investigator — HOSPITAL DE LA SANTA CREU I SANT PAU, Servicio de Oncología Médica; Carmen Garcias de España, MD, Principal Investigator — HOSPITAL UNIVERSITARI SON ESPASES, Servicio de Oncología Médica; Teresa Alonso, MD, Principal Investigator — HOSPITAL RAMÓN Y CAJAL, Servicio de Oncología Médica; Javier Puente, MD, Principal Investigator — HOSPITAL CLÍNICO SAN CARLOS, Servicio de Oncología Médica; Martín Lázaro, Md, Principal Investigator — COMPLEXO HOSPITALARIO UNIVERSITARIO DE VIGO, Servicio de Oncología Médica; Javier Cassinello, MD, Principal Investigator — HOSPITAL UNIVERSITARIO DE GUADALAJARA, Servicio de Oncología Médica; María J Méndez, MD, Principal Investigator — COMPLEJO HOSPITALARIO REGIONAL REINA SOFÍA, Servicio de Oncología Médica; Begoña Perez-Valderrama, MD, Principal Investigator — COMPLEJO HOSPITALARIO REGIONAL VIRGEN DEL ROCIO, Servicio de Oncología Médica
Locations (17):
- Spain (17):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Complejo Hospitalario Regional Reina Sofía, Córdoba
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen de La Victoria, Málaga
  - Complejo Hospitalario Regional Virgen Del Rocio, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Climent MA, Font A, Duran I, Puente J, Jose Mendez-Vidal M, Saez MI, Santander Lobera C, Angel Arranz Arija J, Gonzalez-Del-Alba A, Sanchez-Hernandez A, Juan Fita MJ, Esteban E, Alonso-Gordoa T, Mellado Gonzalez B, Maroto P, Lazaro-Quintela M, Cassinello-Espinosa J, Perez-Valderrama B, Garcias C, Castellano D. A phase II randomised trial of abiraterone acetate plus prednisone in combination with docetaxel or docetaxel plus prednisone after disease progression to abiraterone acetate plus prednisone in patients with metastatic castration-resistant prostate cancer: The ABIDO-SOGUG trial. Eur J Cancer. 2022 Nov;175:110-119. doi: 10.1016/j.ejca.2022.08.002. Epub 2022 Sep 11. PMID 36099670